CLINICAL TRIAL: NCT00868985
Title: Effects of Oral PEG 3350 on the Electrolyte Balance in Patient Volunteers With Chronic Constipation:Pharmacokinetic Evaluation
Brief Title: Effects of Oral PEG 3350 on Electrolyte Balance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Vice President Clinical Development, Norgine Ltd
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PEG-01/2007(ELE)
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Chronic Constipation
MeSH Terms: interventions — polyethylene glycol 3350; Electrolytes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEG 3350 plus electrolytes (Experimental): Patients were dosed with PEG 3350 with electrolytes
  Interventions: Drug: PEG 3350 plus electrolytes
- PEG 3350 without electrolytes (Experimental): Patients were dosed with PEG 3350 without electrolytes
  Interventions: Drug: PEG 3350 without electrolytes

INTERVENTIONS:
Drug: PEG 3350 plus electrolytes — Each patient was treated with PEG 3350 with electrolytes for 10 days at a dose of either one, two or three sachets per day.
  Arms: PEG 3350 plus electrolytes
Drug: PEG 3350 without electrolytes — Each patient was treated with PEG 3350 for 10 days at a dose of either one, two or three sachets per day.
  Arms: PEG 3350 without electrolytes

SUMMARY:
The study is to evaluate the influence of three different doses of PEG 3350 with or without electrolytes on the electrolyte balance in patient volunteers with confirmed chronic constipation.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects written informed consent must be obtained prior to inclusion.
2. Male and female patients between 18 and 70 years of age with confirmed chronic constipation after the run-in period; this is defined as patients who have recorded in their diaries less than 3 bowel motions/week plus one of the following symptoms:

   Straining during at least 25% of defecations Lumpy or hard stools with at least 25% of defecations Sense of incomplete evacuation with at least 25% of defecation Sensation of ano-rectal blockage with at least 25% of defecation Manula manoeuvres of facilitate at least 25% of defecation
3. Willing and able to follow the entire procedure and to comply with the study instructions.
4. For the subgroup of patient volunteers taking ACE-inhibitors (36 subjects): A history of hypertension, with blood pressure controlled to acceptable levels by a stable regimen of ACE-inhibitors.

Exclusion Criteria:

1. Participation in a clinical research study involving investigational drugs or dosage forms within the previous 3 months.
2. Subjects who have previously been enrolled in this study.
3. Subjects who are currently or have a history of abuse of alcohol, non-medical drugs, medicinal drugs or other substance abuse eg solvents.
4. Major surgery in within the last 12 months.
5. Malignant tumors within the last 5 years.
6. Uncontrolled blood pressure or terminal cardiac, liver and/or kidney diseases.
7. Clinical relevant acute gastrointestinal tract disease, including evidence of intestinal perforation or obstruction, paralytic ileus, toxic megacolon, severe inflammatory conditions.
8. Acute urinary tract conditions, including cystitis.
9. Patients with diagnosis or evidence of the following diseases: Hypothyroidism, diabetes mellitus, porphyria, pituitary gland insufficiency, pheochromocytoma, glucagonoma, neurological diseases (eg Hirschprung disease, neurofibromatosis, Chagas disease, stroke, autonomous neuropathy, intestinal pseudoobstruction, Multiple sclerosis, medullar injury, Parkinson disease, Shy-Drager syndrome), collagenosis, vasculitis, myopathy (e.g. sclerodermatitis, amyloidosis, dermatomyositis), intoxication with heavy metals (e.g. Pb, As, Hg)
10. Concomitant medication:

    1. Use of any oral purgatives/laxatives and prokinetics within the last 14 days prior to dosing.
    2. Use of any opioids, anti-cholinergics, tricyclic anti-depressants, MAOIs, Fe preparations, within the 4 weeks prior to dosing.
    3. Use of any Ca-antagonists, Beta-blockers or diuretics within the last 4 weeks prior to dosing.
    4. other medication which in the opinion of the Investigator could interfere with the principal function of the GI tract.
11. Subject unable to provide written consent.
12. Failure to satisfy the Investigator of fitness to participate for any other reason, including suspected non-compliance.
13. Women of childbearing potential, who are not using and not willing to use medically reliable methods of contraception for the entire study duration, unless they are surgically sterilised/hysterectomised or any other criteria considered sufficiently reliable by the Investigator in individual cases.
14. Patients with electrolytes disturbances or clinical signs of dehydration.
15. Positive test at screening for HIV or hepatitis.
16. Any clinically significant abnormal test results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Electrolyte profile in blood, urine and faeces, serum osmolality and effect on the renin/aldosterone ratio | Ten days

SECONDARY OUTCOMES:
Amount of PEG 3350 in plasma, urine and faeces | Ten days

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Jürgen Gruss, MD, Study Director — Norgine; Rodica Cinca, MD, Principal Investigator — IFE Human Pharmacology
Locations (1):
- IFE Human Pharmacology, Timișoara, Romania